CLINICAL TRIAL: NCT06742320
Title: Effect of Education on Asthma Knowledge, Control and Quality of Life in School-Age Children Diagnosed With Asthma
Brief Title: The Effect of Education Given to Children With Asthma
Acronym: RCT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Atiye Yıldırım, specialist nurse, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2024/10-06
Record Dates: First submitted 2024-12-16; First posted 2024-12-19 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Asthma
Keywords: asthma; children; education; randomized control
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Intervention Model Description: The study is an experimental type with a pre-test, post-test and follow-up test control group.
Who Masked: Participant, Outcomes Assessor
Masking Description: Children will be randomly assigned to the training and control groups via a computer program.This process was carried out by a person other than the researchers.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education Group (Experimental): Pre-test forms were applied to the children in the training group face to face by the researchers in the outpatient clinic. Children assigned to the training group received asthma education in a single session, 3 modules/each module lasting at least 15 minutes. Post-test forms were administered immediately after the training.The 2nd and 3rd follow-up tests will be administered online via Google Form in the 1st and 3rd months after the training is completed.
  Interventions: Behavioral: Asthma education
- Control group (No Intervention): Pre-test forms will be applied to the control group face-to-face by researchers in the outpatient clinic.In the control group, follow-up tests (three weeks, 1 month and 3 months after the pre-tests) will be administered online via Google Form.

INTERVENTIONS:
Behavioral: Asthma education — There are very few studies examining the asthma knowledge level, quality of life and asthma control of children in Turkey.
  Arms: Education Group

SUMMARY:
The aim of this study is to examine the effects of asthma education on asthma knowledge, control and quality of life of school-aged children (7-11 years old) diagnosed with asthma and followed up in the outpatient clinic.

DETAILED DESCRIPTION:
Asthma is among the most common chronic diseases in childhood. Besides being one of the most common diseases, it is a preventable and controllable disease.In a study analyzing asthma data of children aged 0-17 by the Centers for Disease Control and Prevention (CDC), the prevalence of asthma was 8.7% in 2001, this rate increased to 9.4% in 2010, and decreased to 8.3% in 2016. In the same study, the prevalence of asthma was found to be 9.2% in boys and 7.4% in girls.Asthma is also the leading cause of school absences in children ages 5 to 17, accounting for more than 14 million days of absence from school in 2013.These adverse effects of asthma can be minimized with appropriate education.Studies have found an increase in the quality of life of asthmatic students after asthma education, a decrease in asthma exacerbations, school absences, parental workday loss and medical expenses, and an increase in adherence to treatment, asthma knowledge and correct inhaler use.These findings suggest that asthma management interventions increase children's knowledge about their disease and their self-management skills.Based on this need, the aim of this study is to examine the effects of asthma education given to school-aged children (7-11 years old) diagnosed with asthma and followed up in the outpatient clinic on their asthma knowledge, control and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 7-11,
* Medically diagnosed with asthma and being followed up in the outpatient clinic
* Family and child agreeing to participate in the study
* Ability to use a smartphone, computer or tablet
* Having internet access
* Children who can read and understand Turkish

Exclusion Criteria:

* Children who do not have a medical diagnosis of asthma
* Children who do not agree to participate in the study and their parents
* Children who do not complete the training and tests

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 72 (Estimated)
Dates: Start 2024-07-25 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2025-03-15 (Estimated)

PRIMARY OUTCOMES:
Asthma Quality of Life Scale for Children | About 3 months
  The scale was developed for children aged 7-11 and adapted to Turkish by Yüksel et al. (2009) and consists of 3 sub-dimensions, namely 'asthma symptoms', 'activity limitation' and 'emotional function', and 23 questions. Scoring varies between 1-7 for each item.The total score to be obtained from the scale is between 23 and 161. A high score indicates a good quality of life.
Childhood Asthma Control Test | About 3 months
  The scale evaluates asthma symptoms in the last 4 weeks for children aged 4-11. Children answer the first 4 questions themselves, while the person responsible for the child's care answers the last 3 questions. The total score to be obtained from the scale is between 0-27. Patients with a total score of 19 points and below are considered to have uncontrolled asthma, and patients with a score of 20 points and above are considered to have controlled asthma.

SECONDARY OUTCOMES:
Asthma Knowledge Survey | About 3 months
  The asthma knowledge survey, which was created by the researchers by reviewing the relevant literature, consists of 13 questions. The first 8 questions in the survey are about asthma definition, symptoms, triggers and physical activity status, and the last 5 questions are about asthma treatment. The questions have a 3-point answer option of yes, no/I don't know. 1 point is received for correct answers and 0 points are received for wrong/I don't know. There is a total distribution between 0-13 points. The survey items were rearranged in line with the opinions received from 9 experts. The content validity rates of the scores given by the experts to the items vary between 0.85-1.0. The content validity index was calculated as 0.98 in the study. It was determined that there was a high level and statistically significant consensus among the experts.

CONTACTS AND LOCATIONS:
Locations (1):
- Dokuz Eylul University Nevvar & Salih İşgören Children's Hospital Pediatric Allergy and Immunology Polyclinic, Izmir, Balcova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
I haven't decided yet.